CLINICAL TRIAL: NCT00321321
Title: Phase 2 Study of The Beta Cell Responsiveness to GIP With and Without Sulfonylurea in Patients With Type 2 Diabetes
Brief Title: The Beta Cell Responsiveness to Glucose-dependent Insulinotropic Polypeptide (GIP) With and Without Sulfonylurea in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Kasper Aaboe, Gentofte University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KA-05011
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Results first posted 2008-10-02 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2008-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Glucose dependent insulinotropic polypeptide; Sulfonylurea compounds; insulin secretion; Sulfonylurea receptor subunit-SUR1; Impaired incretin effect
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sulfonylurea

SUMMARY:
The investigators hypothesize that the impaired insulinotropic effect of the incretin hormone GIP may be due to inadequate sensitization and ATP induced closure of beta cell K-ATP channels. By closing the channels through the use of sulfonylurea (SU) we hope to restore the insulinotropic effect of GIP.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus diagnosed according to WHO criteria
* Diet and/or metformin treatment
* HbA1c > 7,0% for metformin treated patients
* HbA1c > 7,5% for diet treated patients
* Age: 18 years or older
* 25 > BMI > 40 kg/m2
* Signed informed consent
* Sufficient birth control in case of child bearing capacity

Exclusion Criteria:

* Proliferative retinopathy
* Diabetic nephropathy with s-creatinine > 130 microM and/or macroalbuminuria
* Liver disease (ALAT > 2 x normal value)
* CAD (NYHA group III or IV)
* Positive screening for islet-cell and/or GAD-65 autoantibodies
* Type 1 diabetes i first degree relatives
* Gastrointestinal surgery with intestinal resection
* Anemia
* Pregnancy and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Aaboe, M.D., Principal Investigator — Gentofte University Hospital
Locations (1):
- Department of Internal Medicine, Gentofte University Hospital, Hellerup, Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May 2006 - March 2007, Outpatient clinic and advertisement
Period: Overall Study
Arm/Group | Sulfonylurea
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sulfonylurea
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  Denmark | 12

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion
Description: area under the curve AUC and insulin secretion rate
Time Frame: 0 - 90 minutes
Measure: Number; unit: pmol/l * 90 minutes
Arm/Group | Sulfonylurea
Number analyzed (Participants) | 12
pmol/l * 90 minutes | 56766

ADVERSE EVENTS:
Groups:
- Sulfonylurea: Sulfonylurea-treated patients
Arm/Group | Sulfonylurea
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes